CLINICAL TRIAL: NCT05223374
Title: Extension for Community Healthcare Outcomes (ECHO) Autism Diagnostic Study in Primary Care Setting
Status: Completed | Type: Observational
Sponsor: Cognoa, Inc. (Industry)
Collaborators: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: 2075722
Record Dates: First submitted 2022-01-20; First posted 2022-02-04 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2022-01

CONDITIONS: Children18-72 Months With a Suspicion Autistic Disorder
Keywords: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Assess the time to diagnosis from initial concern by EAC utilizing Canvas Dx: Time from initial concern to diagnosis when using Canvas Dx as part of the diagnostic process (Reported time to diagnosis)
  Interventions: Device: Canvas Dx

INTERVENTIONS:
Device: Canvas Dx — Canvas Dx is intended for use by healthcare providers as an aid in the diagnosis of autism spectrum disorder (ASD) for patients ages 18 months through 72 months who are at risk for developmental delay based on concerns of a parent, caregiver, or healthcare provider. The device is not intended for use as a stand-alone diagnostic device but as an adjunct to the diagnostic process. The device is for prescription use only (Rx only)

SUMMARY:
This is a collaborative study that will provide a comprehensive source of observational data that can be used to obtain real world evidence of ASD. The study will contain demographic and observational clinical data for eligible participants. All decisions regarding patient care will be determined by the ECHO Autism Clinician (EAC). All clinical outcomes will be assessed by the EAC as would occur in routine clinical practice.

DETAILED DESCRIPTION:
The study will be conducted by the University of Missouri ECHO Autism Communities Research Team (RT). Research participants recruited by the RT will include: 1) University of Missouri ECHO Autism Community trained clinicians (EACs) in both rural and suburban areas across the United States; 2)Caregivers/Patients with a suspicion of autism. Caregivers/Patients with a suspicion of autism and EACs will complete the informed consent process prior to entering the study. Once enrolled, EACs will provide routine clinical care and conduct best-practice ECHO Autism diagnostic evaluations with the addition of Canvas Dx to patients who have a suspicion of autism spectrum disorder. Canvas Dx will be prescribed; the caregiver will download and access the diagnostic app with a code. The caregiver will then complete the following activities:

* Complete Caregiver Questionnaire in the mobile app
* Upload two 90 sec to 5-minute videos of the participant through the mobile app

ELIGIBILITY:
Inclusion Criteria:

1. English is spoken proficiently by the participating patient/family, in the opinion of the EAC.
2. Meets labeling of device
3. Parent, guardian, or legally authorized representative (LAR) must be able to read, understand, and sign and date the Informed Consent Form (ICF)
4. Sex assigned at birth (Female or male or non-binary)
5. Female or male, > 18 to < 72 months of age
6. Caregiver, HCP or community-based professional concern for developmental delay or Autism
7. Parent/guardian/LAR must have smartphone utilizing the most recent and previous version of iOS and Android operating systems (iOS 13 or 14; Android 10 or 11, excluding Android Go)
8. Participants must be willing to be videotaped as part of the device input

Exclusion Criteria:

1. Participants with a prior diagnosis of Autism Spectrum Disorder (ASD) rendered by a healthcare professional
2. Participants with any other medical, behavioral, or developmental condition that in the opinion of the ECHO Autism Clinician may confound study data/assessments
3. Participants whose age on the date of enrollment is outside the target age range
4. Participants or caregivers who have, to the best of their knowledge, been previously enrolled in any Cognoa clinical study or survey

Ages: 18 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 18-72 months who have a suspicion of ASD.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-02-04 (Actual); Study Completion 2024-02-04 (Actual)

PRIMARY OUTCOMES:
Assess the time to diagnosis from initial concern by EAC utilizing Canvas Dx | up to 2 months
  Assessing the time frame to diagnosis from the initial concern by the EAC utilizing Canvas Dx

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Sohl, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- ECHO Autism, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided
The Clinical Study Report (CSR) findings will be shared once analyzed.

REFERENCES:
- [Derived] Sohl K, Linstead E, Heinz K, Lledo EE, Brewer Curran A, Mahurin M, Nanclares-Nogues V, Salomon C, Seal M, Taraman S. Integration of an Artificial Intelligence-Based Autism Diagnostic Device into the ECHO Autism Primary Care Workflow: Prospective Observational Study. JMIR Form Res. 2025 Oct 21;9:e80733. doi: 10.2196/80733. PMID 41124399
- [Derived] Sohl K, Kilian R, Brewer Curran A, Mahurin M, Nanclares-Nogues V, Liu-Mayo S, Salomon C, Shannon J, Taraman S. Feasibility and Impact of Integrating an Artificial Intelligence-Based Diagnosis Aid for Autism Into the Extension for Community Health Outcomes Autism Primary Care Model: Protocol for a Prospective Observational Study. JMIR Res Protoc. 2022 Jul 19;11(7):e37576. doi: 10.2196/37576. PMID 35852831